CLINICAL TRIAL: NCT02122302
Title: Online Health Assessment to Support Comprehensive Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to unsuccessful accrual.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Los Angeles (Other); Northwestern University (Other); Beth Israel Deaconess Medical Center (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Simon K. Lo, M.D., Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00027150; 1R43DK092097 (NIH)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pancreatitis
Keywords: Altered gastrointestinal anatomy; Chronic pancreatic disease; Chronic pancreatic pain; Patient self-assessment; Online assessment
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Web-based health assessment (Experimental)
  Interventions: Device: CarePrep Online Health Assessment

INTERVENTIONS:
Device: CarePrep Online Health Assessment — Patients can utilize a web-based self-assessment system to answer questions that address medical, psychological, social, behavioral, and quality-of-life issues that are relevant to pancreatic disease. Patients can enter and track their symptoms over the Internet from home or clinic. The system is also designed to gather clues to identify neuropathic pain, which occurs when the nervous system fails to properly regulate pain signals.
  Other Names: Online CarePrep Assessment (OCA)

SUMMARY:
This investigation develops an online, patient self-assessment system, called "CarePrep" to support the care and clinical research of patients with chronic pancreatic disease and chronic pancreatic pain. This web-based assessment presents patients with questions that address medical, psychological, social, behavioral, and quality-of-life issues that are relevant to pancreatic disease. Patients will be given the opportunity to enter and track their symptoms over the Internet from home or clinic. The system is also designed to gather clues to identify neuropathic pain, which occurs when the nervous system fails to properly regulate pain signals. Any of these factors can contribute to chronic pain and may point the way to more effective treatment. The broad objective of this study is to extend CarePrep to cover a full range of topics that are relevant to chronic pancreatic disease. The study team will refine this content based on the system's accuracy in real clinical settings and direct efforts to maximize its feasibility.

DETAILED DESCRIPTION:
The following aims will be addressed:

Aim 1: Refine and extend CarePrep content for targeted disorders.

Working with experts at our sites, the study team will review CarePrep content in association with current literature and established instruments. Applying this data, a comprehensive pain assessment will be developed and content to target chronic pancreatic pain (CPP) will be prioritized. During Phase 1 of the study, the system will be deployed, patient testing begun, and feedback gathered to guide refinement. Patients will be asked to complete their online CarePrep assessment before their scheduled clinic visit; the report will be delivered to their attending physician prior to the clinic encounter. Patients who are unable to complete their assessment at home will have access to electronic tablets which will be provided in clinic.

Aim 2: Test with patients, gather feedback, and conduct cognitive and structured interviews to assess validity.

Research staff will conduct individual patient interviews to assess CarePrep validity, via the following ways: Cognitive interviews probing for CarePrep comprehension and ease of use, as well as measuring patients' rationale for selecting their online responses; structured interviews that will include a block of standardized questions that mirror the online CarePrep assessment (patients' interview responses will be compared to data from their online session to assess the sensitivity of CarePrep screening questions); and patients' ratings of CarePrep's accuracy will be collected to improve and validate system design.

Aim 3: Assess feasibility.

In Phase II of the study, physician and patient self-reports will be used to assess feasibility and utility. The objective of this phase is to deliver a system that supports a comprehensive health assessment and facilitates physician-patient communication so that physicians will adopt the system for routine care.

ELIGIBILITY:
Inclusion Criteria:

* Be a current or future patient of the Cedars-Sinai Medical Center's Pancreaticobiliary clinic
* Read English
* Have access to a computer or touch-screen tablet to complete the online assessment

Exclusion Criteria:

* Patients unable or unwilling to complete the online assessment at home or in clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Physician and patient evaluation of validity and feasibility of online patient self-assessment system to support integrated gastrointestinal and biopsychosocial care | One year
  Feedback via cognitive and structured interviews will assess validity: Cognitive interviews will probe for CarePrep comprehension and ease of use and will measure patients' rationale for selecting their online responses; structured interviews will include a block of standardized questions mirroring the online CarePrep assessment; patients' interview responses will be compared to data from their online session to assess the sensitivity of CarePrep screening questions; patients' ratings of CarePrep's accuracy will be collected to improve and validate system design; and experts and clinicians will review relevant sections of the CarePrep report for accuracy in order to address the utility and accuracy of reported data..
  Physician and patient self-reports will assess feasibility and utility: After the refinement and validation phases have been completed, patients and clinicians will score the usefulness of Careprep in routine clinic use via brief self-reports.

CONTACTS AND LOCATIONS:
Overall Officials: Simon K Lo, M.D., Principal Investigator — Cedars-Sinai Medical Center; Stephen J Pandol, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States